CLINICAL TRIAL: NCT01266382
Title: The Effect of AposTherapy on the Level of Pain, Function and Quality of Life in Patients With Neuro-muscular and Neurological Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Collaborators: Apos Medical and Sports Technology Ltd. (Industry)
Purpose: Treatment
Other Study IDs: 93/09
Record Dates: First submitted 2010-12-22; First posted 2010-12-24 (Estimated); Last update posted 2010-12-24 (Estimated); Status verified 2009-07

CONDITIONS: Osteoarthritis; Spinal Diseases; Ligament Rupture; Lower Extremity Fracture; Neurological Disorders
MeSH Terms: conditions — Osteoarthritis; Spinal Diseases; Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: AposTherapy — a biomechanical device including 2 hemispheric biomechanical elements attached to a platform in a form of a shoe. the biomechanical device is calibrated to each patient by a physiotherapist specialized with the treatment methodology. patient are instructed to walk indoor with the device. time of exercise is gradually increase

SUMMARY:
The purpose of the study is to examine the effect of a new biomechanical device and treatment methodology (AposTherapy) on gait patterns, pain, function and quality of life of patients with musculoskeletal and neurological disorders. Based on previous reports the investigators hypothesis that this therapy will have a positive effect on these measurements.

ELIGIBILITY:
Inclusion Criteria:

* Primary osteoarthritis
* Lower limb joint replacement
* Lower limbs fractures
* Spinal disorders including LBP w/wo refered symptoms, radiculopathy, spinal stenosis
* ligaments tear
* Meniscal tears

Exclusion Criteria:

* lack of balance (3 falls in the last year)
* incapable to complete a questionnaire •>age 85

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Spatio-temporal Gait parameters
WOMAC
SF-36

SECONDARY OUTCOMES:
FAOS questionnaire
Oswestry questionnaire
Clinical measurements

CONTACTS AND LOCATIONS:
Locations (1):
- AposTherapy center, Herzliya, Israel

REFERENCES:
- [Derived] Segal G, Bar-Ziv Y, Velkes S, Benkovich V, Stanger G, Debbi EM, Debi R, Mor A, Elbaz A. A non-invasive biomechanical device and treatment for patients following total hip arthroplasty: results of a 6-month pilot investigation. J Orthop Surg Res. 2013 May 21;8:13. doi: 10.1186/1749-799X-8-13. PMID 23692690